CLINICAL TRIAL: NCT01136239
Title: The Effect of High Dose N-acetylcysteine on Airtrapping and Airway Resistance of Chronic Obstructive Pulmonary disease-a Double Blinded Randomized Placebo Controlled Trial
Brief Title: The Effect of High Dose N-acetylcysteine on Airtrapping and Airway Resistance in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Tse Hoi Nam, Specialist in Respiratory medicine, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KW/EX/09-140; PR/CT 324/2009 (Other: Department of Health, Hong Kong)
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: COPD
Keywords: COPD; N-acetylcysteine; airtrapping; airway resistance; antioxidant
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (600mg twice daily)
  Interventions: Drug: Placebo
- N-acetylcysteine (Active Comparator): N-acetylcysteine (600mg twice daily)
  Interventions: Drug: N-acetycysteine (600mg twice daily)

INTERVENTIONS:
Drug: N-acetycysteine (600mg twice daily) — N-acetycysteine (600mg twice daily) for one year
  Arms: N-acetylcysteine
Drug: Placebo — Placebo (600mg twice daily)
  Arms: Placebo

SUMMARY:
This study is to investigate the add-on effect of high dose NAC (600mg tablet twice daily) on reduction of airtrapping and airway resistance in stable COPD patients as well as to study it's effect in reducing exacerbation, improving exercise capacity and quality of life in stable COPD patients.

DETAILED DESCRIPTION:
Background: The mucolytic and antioxidant effects of N-acetylcysteine (NAC) may be of great value in treatment of COPD patients. However, previous studies fail to demonstrate the beneficial effect of NAC. This may be due to insufficient dose of NAC used as well as inadequate outcome parameters measured in the past studies.

Objective of study: This study is to investigate the add-on effect of high dose NAC (600mg tablet twice daily) on reduction of airtrapping and airway resistance in stable COPD patients as well as to study it's effect in reducing exacerbation, improving exercise capacity and quality of life in stable COPD patients.

Study design: Randomized double blinded placebo controlled trial in Kwong Wah Hospital

Methodology: Patients are recruited in Kwong Wah Hospital if they fulfill the spirometric criteria of COPD. Eligible subjects will be randomized into the treatment (NAC 600mg tablet twice daily) and placebo group after completion of run in period. NAC and placebo will be prescribed accordingly in addition to their usual therapy. Both patients and investigators are blinded about the group allocation. Baseline assessment will be done and patients will be followed up at 16th weeks and 52th week of the study.

During each follow-up visit, hyperinflation parameters like inspiratory capacity (IC) will be measured by plethysmography. Airway resistance will be measured by both plethysmography and impulse oscillometry machine. Exercise capacity (6 min walking distance) and quality of life are also recorded during each follow up.

The difference of the above parameters between the 2 groups (drug and placebo group) will be analyszed by the Repeated measures ANOVA test

ELIGIBILITY:
Inclusion Criteria:

* Spirometry diagnosed COPD with FEV1/FVC ratio less than 70% and FEV1 less than 80% predicted
* clinically stable and exacerbation free in the past 4 weeks
* history of at least one COPD exacerbation in the past one year

Exclusion Criteria:

* patients allergic or intolerant to NAC
* Recent use of NAC in the past one month
* history of asthma, non COPD respiratory disorders like bronchiectasis, pneumoconiosis or any active pulmonary infection
* patients on long term steroid
* patients on long term oxygen therapy or non invasive ventilation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Airtrapping in COPD patients | At baseline (time 0 week)
  The airtrapping of COPD patients is measured by inspiratory capacity (IC), using plethsmography (MedGraphics Elite series)
Airtrapping in COPD patients | At 16th week
  The airtrapping of COPD patients is measured by inspiratory capacity (IC), using plethsmography (MedGraphics Elite series)
Airtrapping in COPD patients | At 52th Week
  The airtrapping of COPD patients is measured by inspiratory capacity (IC), using plethsmography (MedGraphics Elite series)

SECONDARY OUTCOMES:
Airway resistance in COPD patients | At baseline ( time 0)
  Airway resistance is measured by plethsmography (Medgraphics Elite series) and impulse oscillometry.
Airway resistance in COPD patients | At 16th week
  Airway resistance is measured by plethsmography (Medgraphics Elite series) and impulse oscillometry.
Airway resistance in COPD patients | At 52th week
  Airway resistance is measured by plethsmography (Medgraphics Elite series) and impulse oscillometry.
Exercise capacity | At baseline ( time 0)
  Exercise capacity is measured by 6-min-walking distance (6MWD)and it is performed by a trained physiotherapist
Exercise capacity | At 16th week
  Exercise capacity is measured by 6-min-walking distance (6MWD)and it is performed by a trained physiotherapist
Exercise capacity | At 52th week
  Exercise capacity is measured by 6-min-walking distance (6MWD)and it is performed by a trained physiotherapist
Quality of life | At baseline (time 0)
  Quality of life is assessed by using the St Qeorge Respiratory Questionnaire (SQRQ)and it will be performed by a trained physiotherapist
Quality of life | At 16th week
  Quality of life is assessed by using the St Qeorge Respiratory Questionnaire (SQRQ)and it will be performed by a trained physiotherapist
Quality of life | At 52th week
  Quality of life is assessed by using the St Qeorge Respiratory Questionnaire (SQRQ)and it will be performed by a trained physiotherapist
COPD exacerbation rate | At 52th week
  The number of COPD exacerbation (exacerbation was defined as 2 out of 3 of the following criteria; 1.increase in shortness of breath, 2. increase in sputum purulence or 3. increase in sputum volume) will be assessed and documented

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Nam Tse, FHKAM, MBChB, Principal Investigator — Kwong Wah Hospital
Locations (1):
- Medical Department, Hong Kong, China

REFERENCES:
- [Derived] Tse HN, Raiteri L, Wong KY, Ng LY, Yee KS, Tseng CZS. Benefits of high-dose N-acetylcysteine to exacerbation-prone patients with COPD. Chest. 2014 Sep;146(3):611-623. doi: 10.1378/chest.13-2784. PMID 24833327
- [Derived] Tse HN, Raiteri L, Wong KY, Yee KS, Ng LY, Wai KY, Loo CK, Chan MH. High-dose N-acetylcysteine in stable COPD: the 1-year, double-blind, randomized, placebo-controlled HIACE study. Chest. 2013 Jul;144(1):106-118. doi: 10.1378/chest.12-2357. PMID 23348146